CLINICAL TRIAL: NCT07283549
Title: Reducing Loneliness Among Older Adults in Hong Kong by Volunteer-delivered Mindfulness and Behavioral Activation Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Education University of Hong Kong (Other)
Responsible Party: Principal Investigator, Chou Kee Lee, Chair Professor of Social Policy, Education University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2023-2024-0570
Record Dates: First submitted 2025-12-04; First posted 2025-12-16 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Loneliness; Mental Health
Keywords: Loneliness; Older Adults; Mental Health; Volunteers; Psychosocial Interventions
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Tele-BA (Experimental): Behavioral Activation
  Interventions: Behavioral: Tele-BA
- Tele-MF (Experimental): Mindfulness
  Interventions: Behavioral: Tele-MF
- Tele-BF (Active Comparator): Befriending
  Interventions: Other: Tele-BF

INTERVENTIONS:
Behavioral: Tele-BA — Behavioral Activation
  Arms: Tele-BA
Behavioral: Tele-MF — Mindfulness
  Arms: Tele-MF
Other: Tele-BF — Befriending
  Arms: Tele-BF

SUMMARY:
This study aims to recruit and train retirees and young people to be volunteers who will deliver the layperson-delivered, telephone-based behavioral activation and mindfulness intervention to older adults.

DETAILED DESCRIPTION:
Retirees and young people will be recruited, trained, and delivered telephone-based psychosocial interventions to older adults.

ELIGIBILITY:
Inclusion Criteria:

* 65 years older and above

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 251 (Actual)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-07-23 (Actual); Study Completion 2025-07-23 (Actual)

PRIMARY OUTCOMES:
Loneliness | Baseline, 4 weeks, 3 months
  UCLA Loneliness Scale; Each item will be rated from 1=Never to 4=Always. Total scores range from 20 to 80.

SECONDARY OUTCOMES:
Loneliness | Baseline, 4 weeks, 3 months
  De Jong Gierveld Loneliness Scale; Each item will be rated from 1=Yes to 3=No. Total scores range from 0 to 6, with subscale score ranging from 0 to 3.
Anxiety | Baseline, 4 weeks, 3 months
  Hospital Anxiety and Depression Scale; Each item will be rated from 0=Not at all to 3=Most of the time. Total score range from 0 to 42.
Sleep Quality | Baseline, 4 weeks, 3 months
  Sleep Condition Indicator; Each item will be rated from 0 to 4. Total score range from 0 to 32.
Stress | Baseline, 4 weeks, 3 months
  Perceived Stress Scale; Each item will be rated from 0=Never to 4=Very often. Total scores range from 0 to 56.
Well-Being | Baseline, 4 weeks, 3 months
  Psychological Well-Being Scale; Each item will be rated from 1=strongly agree to 7=strongly disagree.

CONTACTS AND LOCATIONS:
Locations (1):
- The Education University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No